CLINICAL TRIAL: NCT06501131
Title: The Impact of Partial Visible Light Spectrum Absence on Pupil Response and Autonomic Nervous System Excitability: A Cross-Over Randomized Controlled Trial
Brief Title: A Self-controlled Study of the Effect of Partial Spectral Absence of Visible Light on the Pupil
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2024KYPJ062
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Full Spectrum
Keywords: myopia,spectrum,vegetative nerve,pupil
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- full spectrum light group (Experimental): Subjects were asked to stay in a resting state for 5 minutes in a dark room, then turn on the full-spectrum light and adapt to the light environment for 5 minutes, and then take measurements for 5 minutes. After wash-out in the dark room for 5 minutes, change the light to ordinary LED lamp and repeat the above test steps for measurement.
  Interventions: Other: full-spectrum light exposure
- ordinary LED light group (Experimental): Subjects were asked to stay in a resting state for 5 minutes in a dark room, then turn on the ordinary LED lamp and adapt to the light environment for 5 minutes, and then take measurements for 5 minutes. After wash-out in the dark room for 5 minutes, change the light to full-spectrum light and repeat the above test steps for measurement.
  Interventions: Other: specific spectrum absence light exposure

INTERVENTIONS:
Other: full-spectrum light exposure — Subjects will stay in a room with full spectrum light for 5 minutes. After 5 minutes wash-out period, altenate to the other arm.
  Arms: full spectrum light group
Other: specific spectrum absence light exposure — Subjects will stay in a room with ordinary LED light for 5 minutes. After 5 minutes wash-out period, altenate to the other arm.
  Arms: ordinary LED light group

SUMMARY:
Previous studies have shown that the spectrum of light influences myopia. LED lights with a partially absent light spectrum increase the risk of myopia progression compared to LEDs with a full spectrum, potentially mediated by the excitability of the parasympathetic nervous system. This study intends to compare pupil size and area, as well as parameters regulated by the autonomic nervous system (such as skin bioelectrical activity and heart rate), between LEDs with a full visible spectrum and LEDs with a partially absent spectrum around 470nm and 730nm. We aim to elucidate the physiological mechanism underlying the effect of light spectrum on pupil changes and myopia.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 7-45 years 2. Able to wear multi-channel physiological measurement devices and cooperate with experimental procedures.

  3. Binocular? spherical power between -0.50 to -5.00 diopters, and cylinder power no more than -1.50 diopters.

  4. Voluntarily participate in this study with informed consent form signed.

Exclusion Criteria:

* 1. History of diseases affecting autonomic nervous system function, such as depression and anxiety.

  2. History of eye diseases such as strabismus, amblyopia, keratitis, and glaucoma, which are unsuitable for eye movement test.

  3. History of major systemic diseases or surgeries such as cranial surgery, myocardial infarction, or stroke.

  4. Systemic medication history that may affect autonomic nervous system function, including but not limited to antidepressants, antihistamines, anticholinergics, antipsychotics, and sedative-hypnotic drugs like diazepam or lorazepam.

  5. Use of eyedrops such as mydriatics or miotics that will affect pupil size. 6. Having difficulty in understanding and cooperating with the trial, such as those with disabilities, communication barriers, or those unable to undertake examinations.

  7. Other contradictions that the physician may consider inappropriate for enrolment.

Ages: 7 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
pupil size | 5 minutes
  The pupil diameter is measured in real-time using the Eyelink Portable Duo eye tracker.

SECONDARY OUTCOMES:
Skin conductance response | 5 minutes
  Rapidly changing and short-duration skin surface potentials measured in real-time using the Biopac MP160 multi-channel physiological recorder.
Respiratory movement | 5 minutes
  The amplitude of respiratory movements measured in real-time using the Biopac MP160 multi-channel physiological recorder.
Pulse pressure waveform | 5 minutes
  The amplitude of respiratory movements measured in real-time using the Biopac MP160 multi-channel physiological recorder.
Spherical equivalent refraction | 5 minutes
  Measured with autorefractor and defined as the sum of spherical power and half of the cylinder power.
Uncorrected visual acuity | 5 minutes
  Visual acuity without refractive correction.
Axial length | 5 minutes
  Uncorrected visual acuity: Visual acuity without refractive correction.
Corneal curvature | 5 minutes
  Anterior corneal curvature measured by the Pentacam corneal topographer